CLINICAL TRIAL: NCT06962241
Title: Effect of Maintenance of Intraoperative Normothermia in Cesarean Section on Thermal Comfort, Serum Cortisol and Apgar Score: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sinem Öztürkler, Lecturer Dr, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 41380
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy
Keywords: PREGNANCY; NORMOTERMIA; APGAR SCORE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warming group (Experimental): When the pregnant women in the experimental group were laid on the operating table, they were heated from the back with a heating pad. The heating pad remained on the pregnant woman's back throughout the cesarean section. The cesarean section took an average of 35 minutes from the first surgical incision to the completion of the incision after spinal/epidural anesthesia.
  Interventions: Other: Warming group
- Control Group (No Intervention): The patients in this group are given routine care practices of the clinic.

INTERVENTIONS:
Other: Warming group — When the pregnant women in the experimental group were laid on the operating table, they were heated from the back with a heating pad. The heating pad remained on the pregnant woman's back throughout the cesarean section. The cesarean section took an average of 35 minutes from the first surgical incision to the completion of the incision after spinal/epidural anesthesia.
  Arms: Warming group

SUMMARY:
Cesarean section is a common method of delivery worldwide today. According to WHO, cesarean section accounts for more than 1 in 5 (21%) of all births, and it is predicted that approximately one-third (29%) of births will be by cesarean section by 2030. Although cesarean section is a vital and life-saving surgery, it can unnecessarily put mothers and babies at risk for short- and long-term health problems when performed without a medical necessity. Unintended perioperative hypothermia, defined as the inadvertent lowering of core temperature below 36°C during surgery, is a well-known complication of anesthesia. Hypothermia can increase the risk of infection by suppressing the immune system, prolonging the recovery process, and triggering postpartum complications. Maintaining maternal body temperature during cesarean section helps reduce postoperative complications, reduce the risk of infection, and accelerate the recovery process. It is also critical for the health of the baby. Keeping the newborn's body temperature stable can help minimize risks such as hypoxia at birth. However, there are increasing studies showing that temperature control is not only limited to maternal health but also has serious effects on the baby after birth. Therefore, it is understood that maintaining body temperature during cesarean section is an important factor in improving the quality of life for both individuals. This article aims to deeply examine the role of temperature control during cesarean section on maternal and fetal health and the benefits of this intervention.

ELIGIBILITY:
Inclusion Criteria:• Being 19 years of age or older pregnant

* Being at least a primary school graduate
* Having an elective cesarean section with spinal/epidural anesthesia
* Being at or above the 38th week of pregnancy
* Being in the ASA I (Normal, healthy person with no disease or systemic problem other than surgical pathology that does not cause a systemic disorder) class
* Not being diagnosed with high-risk pregnancy (such as oligodydroamnios, premature membrane rupture, gestational diabetes mellitus, preeclampsia, fetal tachycardia, nonreactive NST, intrauterine growth retardation)
* Having a body mass index of >19 kg/m2 and <40 kg/m2
* Having a singleton pregnancy
* Having a healthy fetus
* Having a fasting period of 2-6 hours before surgery
* Being normothermic (36-37.5°C) (tympanic measurement) before surgery

Exclusion Criteria: •Having comorbidities that require emergency delivery or accompany it (severe preeclampsia, bleeding placenta previa, abruption placenta, cord prolapse, fetal distress)

* Need for intensive care in the mother or newborn after cesarean section
* Being anemic with a hemoglobin value below 10 g/dl according to the World Health Organization (2001)
* Not having platelet values within the reference values
* Having any disease that will disrupt the bleeding clotting mechanism (hemophilia, liver failure, vitamin K deficiency, etc.)
* Having a body core temperature above 37.5°C and below 36°C on the morning of surgery
* Having malnutrition, thyroid function and other endocrine disorders, Parkinson's, peripheral circulatory disorders, Diabetes Mellitus, heart disease and a history of stroke
* Having any deterioration on the skin surface of the arms and legs (ecchymosis, edema, urticaria, etc.)

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women are eligible to work
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Concerns of pregnant women who are warmed by a heating pad | Questions will be asked half an hour before the caesarean section
  Anxiety of pregnant women warmed with a heating pad will be measured with the Trait Anxiety Inventory (STAI). It is indicated by selecting one of the following options: "(1) None, (2) A Little, (3) A Lot and (4) Completely".

SECONDARY OUTCOMES:
Thermal Comfort of Pregnant Women Warmed with a Heating Pad | will be measured half an hour after the cesarean section
  The Thermal Comfort scale will be used to measure the pregnant women's comfort after the Caesarean section, which was warmed with a heating pad.

OTHER OUTCOMES:
The effect of warming pregnant women with a heating pad on the Apgar scores of their babies | The Apgar score of the baby born after cesarean section will be evaluated at the 1st and 5th minutes.
Effect of heating pad on shivering of pregnant women | will be measured half an hour before and half an hour after the caesarean section
  The heating pad will be measured with the shivering scale in pregnant women. Zero means no shake, while 3 means the worst possible shake.
warming affects serum cortisol level of newborns | After birth, blood will be taken from the umbilical cord and serum cortisol levels will be checked.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munday J, Osborne S, Yates P, Sturgess D, Jones L, Gosden E. Preoperative Warming Versus no Preoperative Warming for Maintenance of Normothermia in Women Receiving Intrathecal Morphine for Cesarean Delivery: A Single-Blinded, Randomized Controlled Trial. Anesth Analg. 2018 Jan;126(1):183-189. doi: 10.1213/ANE.0000000000002026. PMID 28514320